CLINICAL TRIAL: NCT01473329
Title: Structured Diabetes Self-Management Education in Primary Care and Metabolic Control: a Randomized Clinical Trial.
Brief Title: Structured Diabetes Self-Management Education in Primary Care and Metabolic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-464
Record Dates: First submitted 2011-11-04; First posted 2011-11-17 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes
Keywords: diabetes care; diabetes education; diabetes control
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Structured Diabetes education (Experimental): The intervention group received a structured DSME course. The course was composed by weekly 2 hour meetings for five weeks total hours group of 10 patient and reinforcement meetings every 4 months, for one year
  Interventions: Other: Structured Diabetes Education

INTERVENTIONS:
Other: Structured Diabetes Education — The intervention group received a structured DSME course adapted from 15. The course was composed by weekly 2 hour meetings for five weeks total hours group of 10 patient and reinforcement meetings every 4 months, for one year

SUMMARY:
Education is the mainstay of treatment of diabetes mellitus (DM), since it is through her that patients are trained to perform the management of your disease. There is a wide range of educational interventions tested in patients with DM, not having been defined so far a universal template that can be standardized and recognized as effective for all individuals with the disease. The present study aims to evaluate the effect of a group based structured education program, applied by a primary care generalist nurse, on metabolic control of type 2 diabetes mellitus (DM2) patients attending a primary care unit.

DETAILED DESCRIPTION:
Design: This was a single-center, parallel-group, randomized study Setting: One Primary Care Unit named Santa Cecília/Hospital de Clínicas de Porto Alegre Basic Unit of health, in Porto Alegre, Brazil.

Patients: Adult subjects (more than 18 years-old) up to the age of 80 years, with Type 2 diabetes, and with A1c >7%, regularly attending the primary care unit in the previous 6 months before the trial.

Exclusion criteria were: history of active infection (eg. osteomyelitis, pulmonary tuberculosis, AIDS), chronic corticosteroids use, unstable angina or myocardial infarction in the last 3 months, advanced renal disease require dialysis, heart failure (New York Heart Association class III and IV), cirrhosis, alcohol or illicit drug use, dementia, actual pregnancy or lactation, current cancer or any disease that might affect survival in the next 5 years.

Intervention: The intervention group (I) attended a five-week education course and reinforcement meetings every 4 months, for one year. The control group (C) received usual medical care.

Measures: Clinical (age, gender, ethnicity, history of hypertension and BP levels, smoking and physical activity), anthropometrical (weight, height, and waist circumference) and laboratorial data (fasting glucose levels, A1c, and lipid profile) The Diabetes knowledge was estimated by a questionnaire composed by 22 questions addressing the information discussed in the meetings and will be referred as type 2 DM knowledge score. This measures were done at 0, 4, 8 and 12 months End-points: The primary endpoint was changes in HbA1c at 4, 8 and 12 months. Additional analyses were done to evaluate changes in type 2 DM literacy, blood pressure (BP), body mass index (BMI) and lipids.

Statistical Analysis: Student t and chi-square test were used to compare baseline continuous and categorical variables, respectively. Variables with non-normal distribution were log transformed. Global linear model (GLM) for repeated measurements, with Bonferroni post-hoc test, was used to analyze changes in the outcomes during the trial. HbA1c values after the interventions were adjusted to baseline A1c and dosage of insulin at 12 months by ANCOVA. All patients with at least one A1c measurement available after randomization were included in the analyses, regardless if they attended all meetings of the education course or not (intention to treat analysis). A P value <0.05 (two-tailed) was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* adult subjects (more than 18 years-old) up to the age of 80 years,
* with DM2 (ref ADA), and with A1c >7%,
* regularly attending a primary care unit in the previous 6 months

Exclusion Criteria:

* history of active infection (eg. osteomyelitis, pulmonary tuberculosis, AIDS),
* chronic corticosteroids use,
* unstable angina or myocardial infarction in the last 3 months,
* advanced renal disease require dialysis,
* heart failure (New York Heart Association class III and IV),
* cirrhosis,
* alcohol or illicit drug use,
* dementia,
* actual pregnancy or lactation,
* current cancer or any disease that might affect survival in the next 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
HbA1c | 4, 8 and 12 months
  The primary endpoint was changes in HbA1c at 4, 8 and 12 months.

SECONDARY OUTCOMES:
Changes in type 2 DM literacy. | 4, 8 and 12 months
  Additional analyses were done to evaluate changes in type 2 DM literacy.
Changes in blood pressure (BP) | 4, 8 and 12 months
  Knowledge of diabetes was estimated by a questionnaire consisting of 22 knowledge scores DM
Changes in Blood pressure | 4, 8 and 12 months
  The BP was measured twice with a digital sphygmomanometer (OMROM) with the patient in a sitting position, after a 5-min rest and with 1-min interval between measurements. The value registered was the medium between two measures
Changes in body mass index (BMI) | 4,8 and 12 months
  The BMI (weight/height2) was calculated
Changes in Lipids | 4,8 and 12 months
  The measure of fasting plasma total cholesterol, HDL and triglycerides were by enzymatic colorimetric method 20. The Low-density lipoprotein cholesterol (LDL) was calculated by the formula of Friedwald equation (LDL = total cholesterol - HDL + Triglycerides/5).